CLINICAL TRIAL: NCT02308956
Title: Task Sharing for the Care of Severe Mental Disorders in a Low-income Country: a Randomised, Controlled Non-inferiority Trial
Brief Title: Task Sharing for the Care of Severe Mental Disorders in a Low-income Country
Acronym: TaSCS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Cape Town (Other)
Collaborators: Addis Ababa University (Other); King's College London (Other); Johns Hopkins University (Other); Columbia University (Other); Armauer Hansen Research Institute, Ethiopia (Other)
Responsible Party: Principal Investigator, Charlotte Hanlon, Principal Investigator, Addis Ababa University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: NIH-95699 (Ethiopia)
Record Dates: First submitted 2014-12-03; First posted 2014-12-05 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Schizophrenia; Bipolar Disorder; Major Depressive Disorder; Schizoaffective Disorder
Keywords: task sharing; task shifting; community mental health care; primary care; Developing country; Sub-Saharan Africa; non-inferiority trial
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder; Depressive Disorder, Major; Psychotic Disorders | interventions — Primary Health Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Integrated mental health in primary care (Experimental): Participants in the new intervention arm will receive a task sharing model of locally-delivered mental health care integrated into primary healthcare. General health workers (health officers, nurses and community-based health extension workers) will be given brief training using the WHO's mental health Gap Action Programme and ongoing supervision in order to deliver mental health care to people with severe mental disorders.
  Interventions: Behavioral: Integrated mental health in primary care
- Psychiatric nurse-led specialist care (Active Comparator): Participants in the active control arm will receive an established model of centralised, specialist mental health care delivered by psychiatric nurses at an out-patient clinic within Butajira general hospital and supported by outreach from project workers.
  Interventions: Behavioral: Psychiatric nurse-led specialist care

INTERVENTIONS:
Behavioral: Integrated mental health in primary care — A task-shared model of collaborative mental health care integrated into the primary care setting.
  Arms: Integrated mental health in primary care
Behavioral: Psychiatric nurse-led specialist care — A centralised, psychiatric nurse-led, hospital out-patient service with outreach from project outreach workers
  Arms: Psychiatric nurse-led specialist care

SUMMARY:
Task sharing mental health care through integration of mental health into primary health care (PHC) is advocated as a means of narrowing the treatment gap for mental disorders in low-income countries. In Ethiopia, it is estimated that only around 10% of people with severe mental disorders (SMDs) ever receive evidence-based treatment for their condition, largely due to scarcity of specialist mental health services. A task-sharing model of mental health care in PHC would be more affordable and accessible to the majority of persons with SMD who do not currently receive evidence-based mental health care. Furthermore, task sharing mental health care with PHC is about to be scaled up in Ethiopia in line with the National Mental Health Strategy. However, the effectiveness of the task sharing model of mental health care for people with SMD has not been evaluated systematically in a low-income country. In this study we propose to investigate non-inferiority of a task sharing model of mental health care in PHC compared to a less accessible, but more specialist, psychiatric nurse-led model of care. The specialist model of care has been demonstrated to be acceptable and associated with improved clinical outcomes for persons with SMD engaged in the service in Ethiopia thus making this an appropriate comparison model against which to evaluate non-inferiority of the task sharing model.

DETAILED DESCRIPTION:
Background and rationale Task sharing mental health care through integration of mental health into primary health care (PHC) is advocated as a means of narrowing the treatment gap for mental disorders in low-income countries. In Ethiopia, it is estimated that only around 10% of people with severe mental disorders (SMDs) ever receive evidence-based treatment for their condition, largely due to scarcity of specialist mental health services. A task-sharing model of mental health care in PHC would be more affordable and accessible to the majority of persons with SMD who do not currently receive evidence-based mental health care. Furthermore, task sharing mental health care with PHC is about to be scaled up in Ethiopia in line with the National Mental Health Strategy. However, the effectiveness of the task sharing model of mental health care for people with SMD has not been evaluated systematically in a low-income country. In this study we propose to investigate non-inferiority of a task sharing model of mental health care in PHC compared to a less accessible, but more specialist, psychiatric nurse-led model of care. The specialist model of care has been demonstrated to be acceptable and associated with improved clinical outcomes for persons with SMD engaged in the service in Ethiopia thus making this an appropriate comparison model against which to evaluate non-inferiority of the task sharing model.

Methods Setting Meskan and Mareko districts, Gurage Zone, and Silti Zone, Southern Nations, Nationalities and People's Region, Ethiopia.

Design A parallel group, randomized, single-blinded, controlled non-inferiority trial.

Participants Adults (aged between 25 and 65 years) with severe mental disorders (DSM-IV diagnoses of schizophrenia or schizoaffective disorder, bipolar disorder or major depressive disorder) of a severity requiring continuing care who were (1) identified during a population-based survey carried out between 1998 and 2001, and are still under active follow-up, or (2) recruited from Butajira hospital psychiatric outpatient clinic.

Participants will be recruited and randomised in two phases. Phase 1 will include participants who are clinically stable, not pregnant or breastfeeding, not on depot medication and who have no co-morbid substance use or complex medical conditions. After a three month evaluation period, and if no safety or quality issues arise, the study will proceed to Phase 2. Phase 2 will include participants who have more complex needs or are less clinically stable.

New intervention Participants in the new intervention arm will receive a task sharing model of locally-delivered mental health care integrated into PHC. The intervention will be offered for 18 months.

Comparison intervention Participants in the active control arm will receive the established model of specialist mental health care delivered by psychiatric nurses at an out-patient clinic within Butajira general hospital and supported by outreach from project workers.

General objective To determine the acceptability, affordability, effectiveness and sustainability of mental health care for persons with SMD delivered by trained and supervised non-specialist, primary health care workers compared with an existing psychiatric nurse-led service.

Specific objectives For persons suffering from SMD in Butajira, Ethiopia,

1. To determine the effectiveness and cost-effectiveness of task sharing mental health care with PHC, compared to psychiatric nurse-led mental health care, on the primary outcome measure of symptom severity and on a series of secondary outcome measures.
2. To examine factors influencing the implementation of the task sharing intervention and future scale up, by examining feasibility, sustainability, quality, and safety, and by qualitative exploration of the experience of task sharing from the perspectives of both PHC workers and patients.

Hypothesis Persons with SMD who receive mental health care task-shared with PHC will have a non-inferior clinical outcome, defined as a difference in the mean symptom score on the Brief Psychiatric Rating Scale, expanded version (BPRS-E), of no more than six points higher, compared to persons with SMD who receive a psychiatric nurse-led model of mental health care, after 12 months of care under the comparison service models.

Sample size A total of 324 participants (162 in each arm) will be required to detect a six point higher mean BPRS-E score in the new intervention arm compared to the active control arm, at 90% power and 95% confidence, allowing for 30% refusals and loss to follow-up (n = 124 for Phase 1 and n = 200 for Phase 2).

Randomisation Sequence generation: Computerized generation of randomization list. Blocked randomization stratified by health centre catchment area.

Allocation concealment: Labelled, sealed envelopes containing cards with intervention allocation administered by an independent clinician.

Implementation: Enrollment will occur after participants have been screened for eligibility, given informed consent (or permission given by guardian) and undergone baseline evaluation. After enrollment, an independent clinician will inform the participant of their allocation status.

Concealment Partial concealment. Outcome assessment and data analysis will be carried out by investigators who are masked to the intervention allocation of participants.

Statistical methods Intention to treat will be the primary approach to data analysis, but per protocol analyses will also be used as this is thought to more conservative in the case of non-inferiority trials. The primary outcome measure will be analysed using linear regression adjusting for baseline symptom severity measured using BPRS-E.

ELIGIBILITY:
Inclusion criteria for phase 1

* Participant in the ongoing Butajira SMD cohort study (at baseline (between 1998 and 2001), cohort participants were aged between 15 and 49 years, resident in the area for at least six months and had a DSM-IV (SCAN) diagnosis of schizophrenia or schizoaffective disorder, bipolar disorder or major depressive disorder)
* Ongoing need for continuing mental health care due to:

  1. being on psychotropic medication at assessment or,
  2. not on medication but symptomatic at the time of assessment, or
  3. have experienced partial or full relapse within the two years preceding the assessment
* Stable clinical condition: either in remission from SMD or with residual symptoms that have been stable over the preceding three months.
* Planning to stay resident in the area for 18 months.
* Able to communicate in Amharic, the official language of Ethiopia.
* Willing to be randomised to either of the service models as described in the protocol.
* Has capacity to consent to participation or permission given by guardian and not refusing to participate
* Resident in catchment area of TaSCS health centres (excluding Butajira health centre)

Exclusion criteria for phase 1

* Suicide attempt within the preceding three months
* Current active suicide intent
* Prescribed Thioridazine, Valproate, Lithium or second generation antipsychotic medications (Risperidone and Olanzapine), as these medications are not be available in psychiatric nurse-led units or PHC settings in Ethiopia. Within the Butajira SMD cohort, only people who have received care from psychiatrist-led units in the capital city, Addis Ababa, might be receiving these medications. At present, fewer than 10 patients are known to be taking one of these medications.
* Prescribed depot medication
* Complex or unstable medical condition interfering with management of psychiatric disorder or requiring ongoing medical treatment from Butajira hospital
* Alcohol or khat dependence or abuse within the last 12 months
* Pregnant or breast-feeding
* Restrained at home
* Refusing to participate in the study

Inclusion criteria for Phase 2 As for Phase 1, but if we are unable to recruit enough participants from the existing Butajira SMD cohort then we will expand recruitment to people with SMD attending the psychiatric out-patient clinic at Butajira hospital. A semi-structured diagnostic interview will be carried out to determine diagnostic eligibility (DSM-IV diagnosis of schizophrenia or schizoaffective disorder, bipolar disorder or major depressive disorder). For participants recruited from Butajira hospital psychiatric out-patient clinic, the minimum age will be 25 years and the participants should have had their first contact with specialist mental health services at least two years prior to recruitment into the trial to ensure comparability with the Butajira SMD cohort sample.

Exclusion criteria for Phase 2

* Current active suicide intent
* Prescribed Thioridazine, Valproate, Lithium or second generation antipsychotic medications (Risperidone and Olanzapine).
* Pregnant or breast-feeding and prescribed depot
* Refusing to participate in the study
* Medical condition requiring ongoing medical treatment from Butajira hospital

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2015-03; Primary Completion 2017-05-16 (Actual); Study Completion 2017-11-16 (Actual)

PRIMARY OUTCOMES:
Brief Psychiatric Rating Scale, Expanded Version (BPRS-E) | 12 months post-randomisation (18 months for secondary outcome)
  Symptom severity scale. Non-inferiority of the experimental intervention is defined as less than six point difference in BPRS-E score between the two arms.

SECONDARY OUTCOMES:
WHO Disability Assessment Scale, version 2.0 (WHODAS 2.0) | 12 and 18 months post-randomisation
  Generic disability scale.
Local functioning scale (disability scale for people with severe mental disorders developed specifically for this trial) | 12 and 18 months post-randomisation
  Contextually appropriate l.
Relapse of mental disorder (Measured using the Life Chart Schedule) | 12 and 18 months post-randomisation
  Measured using the Life Chart Schedule
Patient service satisfaction (Newly developed 'mental health service satisfaction scale' and qualitative interviews.) | 12 and 18 months post-randomisation
  Newly developed 'mental health service satisfaction scale' and qualitative interviews.
Nutritional status (Body mass index.) | 12 and 18 months post-randomisation
  Body mass index.
Service use for physical health care (Client Service Receipt Inventory) | 12 and 18 months post-randomisation
  Captured through reimbursement mechanisms and the Client Service Receipt Inventory
Medication side effects (Antipsychotic Side effect Checklist) | 12 and 18 months post-randomisation
  Measured using the Antipsychotic Side effect Checklist
Patient adherence and engagement (Medication Adherence Measure and tracking of appointment attendance.) | 12 and 18 months post-randomisation
  Medication Adherence Measure and tracking of appointment attendance.
Stigma (Family Interview Schedule (caregivers) | 12 and 18 months post-randomisation
  Internalised stigma of mental illness (patients) and the Family Interview Schedule (caregivers)
Restraint (Proportion chained, restrained of confined in the past month.) | 12 and 18 months post-randomisation
  Proportion chained, restrained of confined in the past month.
Adverse event | 12 and 18 months post-randomisation
  Life Chart Schedule and tracking of serious adverse events.
Quality of clinical care (WHO's mental health gap intervention guide) | 12 and 18 months post-randomisation
  Systematic evaluation of quality of documented care compared to evidence-based recommendations in WHO's mental health gap intervention guide.
Acceptability and feasibility (in-depth interviews with patients, caregivers and health care providers.) | 6 months post-randomisation onwards
  Qualitative study using in-depth interviews with patients, caregivers and health care providers.

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Hanlon, BM BS, PhD, Principal Investigator — Addis Ababa University and King's College London
Locations (1):
- Butajira mental health research office, Butajīra, Ethiopia

REFERENCES:
- [Background] Alem A, Kebede D, Fekadu A, Shibre T, Fekadu D, Beyero T, Medhin G, Negash A, Kullgren G. Clinical course and outcome of schizophrenia in a predominantly treatment-naive cohort in rural Ethiopia. Schizophr Bull. 2009 May;35(3):646-54. doi: 10.1093/schbul/sbn029. Epub 2008 Apr 29. PMID 18448478
- [Background] Federal Democratic Republic of Ethiopia Ministry of Health (2012). National Mental Health Strategy, 2012/13-2015/16. Addis Ababa, Ministry of Health.
- [Background] mhGAP: Mental Health Gap Action Programme: Scaling Up Care for Mental, Neurological and Substance Use Disorders. Geneva: World Health Organization; 2008. Available from http://www.ncbi.nlm.nih.gov/books/NBK310851/ PMID 26290926
- [Background] Overall, J. and D. Gorham (1962). The Brief Psychiatric Rating Scale. Psychological Reports 10: 799-812.
- [Derived] Hanlon C, Medhin G, Dewey ME, Prince M, Assefa E, Shibre T, Ejigu DA, Negussie H, Timothewos S, Schneider M, Thornicroft G, Wissow L, Susser E, Lund C, Fekadu A, Alem A. Efficacy and cost-effectiveness of task-shared care for people with severe mental disorders in Ethiopia (TaSCS): a single-blind, randomised, controlled, phase 3 non-inferiority trial. Lancet Psychiatry. 2022 Jan;9(1):59-71. doi: 10.1016/S2215-0366(21)00384-9. PMID 34921796
- [Derived] Hanlon C, Alem A, Medhin G, Shibre T, Ejigu DA, Negussie H, Dewey M, Wissow L, Prince M, Susser E, Lund C, Fekadu A. Task sharing for the care of severe mental disorders in a low-income country (TaSCS): study protocol for a randomised, controlled, non-inferiority trial. Trials. 2016 Feb 11;17:76. doi: 10.1186/s13063-016-1191-x. PMID 26865254